CLINICAL TRIAL: NCT04332965
Title: The Effect of Non-Surgical Periodontal Treatment on Gingival Crevicular Fluid Periostin Levels in Patients With Gingivitis and Chronic Periodontitis
Brief Title: Periostin and Non-Surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ebru Olgun Erdemir, Professor, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/43
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Periodontal Diseases
Keywords: Chronic periodontitis; Gingival crevicular fluid; Gingivitis; Non-surgical periodontal treatment; Periostin
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis; Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with chronic periodontitis (Experimental): Patients with CP (n=30) had teeth with 30% periodontal bone loss and ≥ 2 non-adjacent sites per quadrant with probing depth (PD) ≥ 5 mm and bleeding on probing.
  Interventions: Procedure: Non-Surgical Periodontal Treatment
- Patients with gingivitis (Experimental): Participants with G (n=30) had gingival index ≥ 2 and other inflammation signs.
  Interventions: Procedure: Non-Surgical Periodontal Treatment
- Participants with periodontal healthy (No Intervention): The H group (n=30) consisted of individuals with no attachment loss, no history of periodontal disease, PD ≤3 mm, and whole-mouth bleeding scores <10%.

INTERVENTIONS:
Procedure: Non-Surgical Periodontal Treatment — Scaling and root planing and polishing with specific curettes were performed to patients and oral hygiene education was provided to each patient.
  Other Names: Initial periodontal therapy
  Arms: Patients with chronic periodontitis; Patients with gingivitis

SUMMARY:
A total of 90 subjects, 30 patients with chronic periodontitis, 30 with gingivitis and 30 periodontally healthy subjects were included. Patients with periodontal disease received non-surgical periodontal treatment. Gingival crevicular fluid periostin levels were assessed at baseline, at the 6th week and the 3rd month after treatment.

DETAILED DESCRIPTION:
Periostin is commonly found in collagen-rich tissues, which is thought to affect the production of collagen fibers. Additionally, periostin is synthesized in tissues exposed to constant mechanical forces such as the periosteum, periodontal ligament, tendon, heart valve and skin. Periostin mediates inflammation and fibrosis during diseases of various organs, including the heart, lung, kidney, skin, liver, skeletal muscle and retina.

This study evaluated periostin levels in gingival crevicular fluid from patients with chronic periodontitis, gingivitis and periodontally healthy as well as the effect of non-surgical periodontal treatment on gingival crevicular fluid periostin levels.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic periodontitis
* Clinical diagnosis of gingivitis
* Clinical diagnosis of periodontal health

Exclusion Criteria:

* have any systemic disease
* to be alcohol consumer
* to receive any periodontal therapy in the past 6 months
* to take any drugs regularly
* to be pregnant and/or lactate

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in periostin | Baseline, 6th week and 3rd month
  Total amount of Periostin (pg/30 sec) in gingival crevicular fluid

SECONDARY OUTCOMES:
Change in periodontal clinical parameter | Baseline, 6th week and 3rd month
  Clinical attachment level (mm) (from cemento-enamel junction to the base of periodontal pocket)